CLINICAL TRIAL: NCT02593682
Title: The Role of Orexin in Human Panic Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2015078
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Results first posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suvorexant Group (Experimental): In this arm, subjects will receive 10 mg suvorexant 2 hours before a one-minute 35% CO2 challenge.
  Interventions: Drug: suvorexant
- Placebo Group (Placebo Comparator): In this arm, subjects will receive a placebo, compounded to look identical to the study drug, 2 hours before a one-minute 35% CO2 challenge.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: suvorexant
  Arms: Suvorexant Group
Drug: placebo
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to provide some information (pilot data) about whether the study drug, suvorexant, (1) affects levels of orexin in people with panic disorder, and (2) is associated with decreased panic symptoms in response to a carbon dioxide (CO2) challenge.

DETAILED DESCRIPTION:
Orexins

Hypocretins (orexins), a more recently identified class of pro-arousal neuropeptides, are synthesized by neurons in the lateral and posterior hypothalamus The main described orexins, orexin A (ORX A) and orexin B (ORX B), are both cleaved from a common precursor peptide, prepro-orexin. Orexin A, a 33 amino-acid residue peptide, appears to be conserved across many mammalian species. Orexin B contains 28 amino acids. Orexins promote a variety of behaviors including alertness, vigilance, locomotion, fight-flight responses, and feeding. The physiological effects of the orexins are mediated via 2 G-protein coupled receptors, ORX1 and ORX2. Orexin A binds with greater affinity to the ORX1 receptor, while orexin A and B bind with similar affinity to the ORX2 receptor.

Orexins and Animal Fear Models

Orexins have been implicated in anxiogenesis in some animal fear models. For example, central (icv) injection of orexin A in mice induced anxiety-like responses in the light-dark exploration test and elevated plus maze.

Using an established, γ-aminobutyric acid (GABA)-deficit, rodent model of panic-vulnerability, the investigators' Indiana University preclinical anxiety collaborators provoked a panic-like response in rodents with an anxiogenic sodium lactate (NaLac) infusion, which response was blunted following either site-specific orexin (ORX) gene silencing or systemic pretreatment with an ORX1 antagonist.

In addition, ORX neurons (peptidergic neurons in the lateral hypothalamus) were shown, in turn, to stimulate discrete efferent sites within an emotional network (e.g., bed nucleus of the stria terminalis) to elicit specific behavioral components of the panic-response following sodium lactate. Taken together, these results support the concept that ORX hypersecretion or ORX neuronal overactivity could also be present in human panic disorder (PD).

Orexins' Emerging Role in Human Anxiogenesis / Panicogenesis

Similar to the NaLac model animals, humans with PD have been reported to have cortical and subcortical GABA deficits. If these GABA deficits also extend to impairment of GABAergic inhibition of dorsomedial hypothalamus (DMH) ORX neurons in PD patients, as predicted by the NaLac animal model, they may result in ORX hypersecretion, increased sympathetic activation, and panicogenesis.

There have been few clinical studies of ORX metabolism or function in human anxiety populations. However, recently generated human pilot data in the principal investigator's (PI's) lab, studying the effects of a well-documented anxiogenic stimulus (35% CO2 inhalation) on behavioral, physiological, and biochemical (plasma ORX A; assayed by a standard radioimmunoassays [RIA] kit) measures, in 1 PD patient and 2 healthy volunteers. In this paradigm, the PD patient had a mild panic episode associated with marked early elevations in plasma ORX levels, relative to the volunteers who had minimal anxiety, consistent with a role for ORX in the initiation or elaboration of the human panic response.

It was also demonstrated that, in contrast to human subjects without any axis I psychiatric disorder or with depression alone without panic, only subjects who had high panic scores but no depression had significantly elevated ORX levels in the cerebrospinal fluid (CSF).

The ORX hyperactivity hypothesis of panic that has been evinced from this work is highly innovative, and promises to broaden the understanding of the neurobiology of human panic disorder, as well as provide new treatment directions.

While there are limitations with using plasma ORX A as a measure of central nervous system (CNS) ORX function, one research group has recently published human data indicating that resting state CSF and plasma ORX A levels are highly correlated.

Accordingly, the central hypothesis of this translational human pilot project, and a more definitive project based on it, is as follows: PD is a human anxiety disorder associated with specific cortical and subcortical GABA deficits that result in disruption of normal inhibitory regulation of pro-arousal ORX neurons. This disruption promotes excessive ORX release, sympathetic activation, and vulnerability to spontaneous or chemically induced panic. Pretreatment with an ORX1 receptor antagonist prior to chemical challenge is therefore expected to block the evoked panic response.

Rationale for the Use of CO2 Inhalation

The 35% CO2 challenge is well documented in the literature as being reliable, safe, and easy to administer. The procedure has acceptable test-retest reliability, and may be used to monitor improvement in clinical status following the administration of antipanic medications.

Approximately 70% of PD patients will have a panic attack in response to this challenge, which closely resembles a real-life panic. Therefore, in addition to resting/baseline measurement of plasma ORX A, CO2-evoked levels of plasma ORX A in PD patients will also be examined, and these responses will be correlated with other behavioral and physiological parameters recorded during the CO2 test. The PI has had considerable experience using PD challenge paradigms in clinical research contexts, and he is very familiar with the application of the 35% CO2 challenge.

Project Aims and Expected Results

The project is a study that gathers pilot data relating to the role of orexin in human panic disorder. The effect sizes generated from this pilot work will permit planning and powering of a larger-scale study. It is anticipated that the study will be completed over the course of one year.

Specific Aim 1 will be to provide a preliminary demonstration that acute administration of the first-in-class, FDA-approved insomnia agent, suvorexant, a mixed ORX1/2 receptor antagonist, will block 35% CO2-induced panic symptoms in PD patients, via amelioration of central ORX neuronal hyperactivity (as reflected in blunted plasma ORX responses to CO2 challenge).

To address Specific Aim 1, a prospective, parallel-group, repeated-measures design will be used to compare behavioral, physiological, and biochemical (plasma ORX) responses in 2 independent, unmedicated groups of PD outpatients (n=6 in each group) at baseline/resting state and after panic provocation due to brief (1 minute) inhalation of a 35% CO2 / 65% O2 gas mixture. PD patients will be randomized, in a double-blind manner, to receive either a single, oral dose of the mixed ORX1/2 receptor antagonist, suvorexant (10 mg dose), or identical placebo, 120 minutes before CO2 challenge.

Expected results: It is expected that, compared to placebo, suvorexant pretreatment will blunt behavioral, physiological, and biochemical (plasma ORX) responses to 35% CO2 in PD, due to suppression of CNS ORX hyperactivity. The effect sizes generated from the pilot work will permit planning and powering of a larger-scale study, to definitively address Specific Aim 1.

ELIGIBILITY:
Inclusion Criteria:

* They must be in stable physical health as determined by a medical evaluation, including physical examination, electrocardiogram, laboratory findings (comprehensive metabolic panel, complete blood count [CBC], free T4, urine pregnancy test, urinalysis), urine toxicology screen, and a negative urine pregnancy test in women of child-bearing potential.
* They must satisfy the new clinical criteria in the Diagnostic and Statistical Manual for Mental Disorders, 5th edition (DSM-5) for a current principal diagnosis of PD as confirmed by a semi-structured, diagnostic interview, the Mini International Neuropsychiatric Interview (MINI), administered by the PI.
* Since clinical depression (MDD) is associated with CSF ORX abnormalities, only patients with a current PD without MDD will be enrolled. They will also be required to have a current Montgomery-Asberg Depression Rating Scale (MADRS) total score <12.
* They will be off all regular psychiatric medications and avoid drinking grapefruit juice for at least 2 weeks prior to the 35% CO2 test.
* They must not be pregnant or breastfeeding a baby; and women of childbearing potential must be using birth control while on this study.

Exclusion Criteria:

* any history of a psychotic disorder, bipolar disorder, MDD, depression not otherwise specified (NOS), obsessive compulsive disorder, an eating disorder, post-traumatic stress disorder, or generalized anxiety disorder
* medical conditions for which suvorexant could be contraindicated, such as narcolepsy
* any other sleep disorder
* a substance use disorder, as defined by the DSM-5, within 6 months of the screening visit
* ongoing use of psychiatric medications in the 2 weeks prior to the 35% CO2 test
* current use of certain drugs, including

  * strong cytochrome P450 3A (CYP3A) inhibitors (such as ketoconazole, itraconazole, posaconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, boceprevir, telaprevir, telithromycin, and conivaptan);
  * moderate CYP3A inhibitors (such as amprenavir, aprepitant, atazanavir, ciprofloxacin, diltiazem, erythromycin, fluconazole, fosamprenavir, imatinib, verapamil);
  * strong CYP3A inducers (such as rifampin, carbamazepine and phenytoin);
  * digoxin
* history of any neurological disorder affecting the CNS
* history of uncontrolled or serious medical illness
* a history of hypersensitivity or allergy to suvorexant
* pregnancy or lactation status, or unwillingness to use birth control while on this study, for women of child-bearing potential
* compromised lung function (e.g., chronic obstructive pulmonary disease [COPD], emphysema, idiopathic pulmonary fibrosis, lung cancer)
* inability to fast the required amount of time prior to study visit 2
* a positive test for cannabinoids, opiates, benzodiazepines, amphetamines, cocaine and metabolites
* out-of-range lab values
* an abnormal EKG
* a score > 12 on the Montgomery-Asberg Depression Rating Scale (MADRS)
* inability or unwillingness to avoid drinking grapefruit juice for two weeks prior to the 35% CO2 challenge test
* a history of sudden onset of muscle weakness (cataplexy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Goddard, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Fresno Medical Education Program, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Lecea L, Sutcliffe JG. The hypocretins/orexins: novel hypothalamic neuropeptides involved in different physiological systems. Cell Mol Life Sci. 1999 Oct 30;56(5-6):473-80. doi: 10.1007/s000180050446. PMID 11212299
- [Background] Sakurai T. The neural circuit of orexin (hypocretin): maintaining sleep and wakefulness. Nat Rev Neurosci. 2007 Mar;8(3):171-81. doi: 10.1038/nrn2092. Epub 2007 Feb 14. PMID 17299454
- [Background] Kato H, Hosoda H, Fukuda T, Masushige S, Kida S. Characterization of the promoter of the mouse preproorexin gene. Biosci Biotechnol Biochem. 2007 Mar;71(3):840-3. doi: 10.1271/bbb.60100. Epub 2007 Mar 7. PMID 17341811
- [Background] Samson WK, et al. Both type 1 and type 2 receptors transmit the behavioral effects of orexin/hypocretin. The FASEB Journal. 2007;21(5):A462.
- [Background] Shekhar A, Keim SR, Simon JR, McBride WJ. Dorsomedial hypothalamic GABA dysfunction produces physiological arousal following sodium lactate infusions. Pharmacol Biochem Behav. 1996 Oct;55(2):249-56. doi: 10.1016/s0091-3057(96)00077-9. PMID 8951961
- [Background] Johnson PL, Truitt WA, Fitz SD, Lowry CA, Shekhar A. Neural pathways underlying lactate-induced panic. Neuropsychopharmacology. 2008 Aug;33(9):2093-107. doi: 10.1038/sj.npp.1301621. Epub 2007 Dec 5. PMID 18059441
- [Background] Johnson PL, Truitt W, Fitz SD, Minick PE, Dietrich A, Sanghani S, Traskman-Bendz L, Goddard AW, Brundin L, Shekhar A. A key role for orexin in panic anxiety. Nat Med. 2010 Jan;16(1):111-5. doi: 10.1038/nm.2075. Epub 2009 Dec 27. PMID 20037593
- [Background] Goddard AW, Mason GF, Almai A, Rothman DL, Behar KL, Petroff OA, Charney DS, Krystal JH. Reductions in occipital cortex GABA levels in panic disorder detected with 1h-magnetic resonance spectroscopy. Arch Gen Psychiatry. 2001 Jun;58(6):556-61. doi: 10.1001/archpsyc.58.6.556. PMID 11386984
- [Background] Deadwyler SA, Porrino L, Siegel JM, Hampson RE. Systemic and nasal delivery of orexin-A (Hypocretin-1) reduces the effects of sleep deprivation on cognitive performance in nonhuman primates. J Neurosci. 2007 Dec 26;27(52):14239-47. doi: 10.1523/JNEUROSCI.3878-07.2007. PMID 18160631
- [Background] Shin YW, Dzemidzic M, Jo HJ, Long Z, Medlock C, Dydak U, Goddard AW. Increased resting-state functional connectivity between the anterior cingulate cortex and the precuneus in panic disorder: resting-state connectivity in panic disorder. J Affect Disord. 2013 Sep 25;150(3):1091-5. doi: 10.1016/j.jad.2013.04.026. Epub 2013 May 17. PMID 23688914
- [Background] Long Z, Medlock C, Dzemidzic M, Shin YW, Goddard AW, Dydak U. Decreased GABA levels in anterior cingulate cortex/medial prefrontal cortex in panic disorder. Prog Neuropsychopharmacol Biol Psychiatry. 2013 Jul 1;44:131-5. doi: 10.1016/j.pnpbp.2013.01.020. Epub 2013 Feb 4. PMID 23391588
- [Background] Strawn JR, Pyne-Geithman GJ, Ekhator NN, Horn PS, Uhde TW, Shutter LA, Baker DG, Geracioti TD Jr. Low cerebrospinal fluid and plasma orexin-A (hypocretin-1) concentrations in combat-related posttraumatic stress disorder. Psychoneuroendocrinology. 2010 Aug;35(7):1001-7. doi: 10.1016/j.psyneuen.2010.01.001. Epub 2010 Feb 8. PMID 20116928
- [Background] Goddard AW, Ball SG, Martinez J, Robinson MJ, Yang CR, Russell JM, Shekhar A. Current perspectives of the roles of the central norepinephrine system in anxiety and depression. Depress Anxiety. 2010 Apr;27(4):339-50. doi: 10.1002/da.20642. PMID 19960531
- [Background] Bonaventure P, Yun S, Johnson PL, Shekhar A, Fitz SD, Shireman BT, Lebold TP, Nepomuceno D, Lord B, Wennerholm M, Shelton J, Carruthers N, Lovenberg T, Dugovic C. A selective orexin-1 receptor antagonist attenuates stress-induced hyperarousal without hypnotic effects. J Pharmacol Exp Ther. 2015 Mar;352(3):590-601. doi: 10.1124/jpet.114.220392. Epub 2015 Jan 12. PMID 25583879
- [Background] Papp LA, Klein DF, Martinez J, Schneier F, Cole R, Liebowitz MR, Hollander E, Fyer AJ, Jordan F, Gorman JM. Diagnostic and substance specificity of carbon-dioxide-induced panic. Am J Psychiatry. 1993 Feb;150(2):250-7. doi: 10.1176/ajp.150.2.250. PMID 8123056
- [Background] Perna G, Barbini B, Cocchi S, Bertani A, Gasperini M. 35% CO2 challenge in panic and mood disorders. J Affect Disord. 1995 Mar 14;33(3):189-94. doi: 10.1016/0165-0327(94)00088-q. PMID 7790671
- [Background] Coryell W, Arndt S. The 35% CO2 inhalation procedure: test-retest reliability. Biol Psychiatry. 1999 Apr 1;45(7):923-7. doi: 10.1016/s0006-3223(98)00241-8. PMID 10202581
- [Background] Bertani A, Caldirola D, Bussi R, Bellodi L, Perna G. The 35% CO2 hyperreactivity and clinical symptomatology in patients with panic disorder after 1 week of treatment with citalopram: an open study. J Clin Psychopharmacol. 2001 Jun;21(3):262-7. doi: 10.1097/00004714-200106000-00003. PMID 11386488
- [Background] van Beek N, Griez E. Reactivity to a 35% CO2 challenge in healthy first-degree relatives of patients with panic disorder. Biol Psychiatry. 2000 May 1;47(9):830-5. doi: 10.1016/s0006-3223(99)00265-6. PMID 10812042
- [Background] Schoepp DD, Wright RA, Levine LR, Gaydos B, Potter WZ. LY354740, an mGlu2/3 receptor agonist as a novel approach to treat anxiety/stress. Stress. 2003 Sep;6(3):189-97. doi: 10.1080/1025389031000146773. PMID 13129812
- [Background] Levine L, Gaydos B, Sheehan D, et al. The mGlu2/3 receptor agonist, LY354740, reduces panic anxiety induced by a CO2 challenge in patients diagnosed wityh panic disorder. Neuropharmacology. 2002;43(2):294.
- [Background] Michelson D, Snyder E, Paradis E, Chengan-Liu M, Snavely DB, Hutzelmann J, Walsh JK, Krystal AD, Benca RM, Cohn M, Lines C, Roth T, Herring WJ. Safety and efficacy of suvorexant during 1-year treatment of insomnia with subsequent abrupt treatment discontinuation: a phase 3 randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2014 May;13(5):461-71. doi: 10.1016/S1474-4422(14)70053-5. Epub 2014 Mar 27. PMID 24680372
- [Background] Salomon RM, Ripley B, Kennedy JS, Johnson B, Schmidt D, Zeitzer JM, Nishino S, Mignot E. Diurnal variation of cerebrospinal fluid hypocretin-1 (Orexin-A) levels in control and depressed subjects. Biol Psychiatry. 2003 Jul 15;54(2):96-104. doi: 10.1016/s0006-3223(02)01740-7. PMID 12873798
- [Background] Kessler RC, McGonagle KA, Zhao S, Nelson CB, Hughes M, Eshleman S, Wittchen HU, Kendler KS. Lifetime and 12-month prevalence of DSM-III-R psychiatric disorders in the United States. Results from the National Comorbidity Survey. Arch Gen Psychiatry. 1994 Jan;51(1):8-19. doi: 10.1001/archpsyc.1994.03950010008002. PMID 8279933
- [Background] Weissman MM, Bland RC, Canino GJ, Faravelli C, Greenwald S, Hwu HG, Joyce PR, Karam EG, Lee CK, Lellouch J, Lepine JP, Newman SC, Oakley-Browne MA, Rubio-Stipec M, Wells JE, Wickramaratne PJ, Wittchen HU, Yeh EK. The cross-national epidemiology of panic disorder. Arch Gen Psychiatry. 1997 Apr;54(4):305-9. doi: 10.1001/archpsyc.1997.01830160021003. PMID 9107146
- [Background] Pollack MH, Otto MW, Rosenbaum JF, Sachs GS, O'Neil C, Asher R, Meltzer-Brody S. Longitudinal course of panic disorder: findings from the Massachusetts General Hospital Naturalistic Study. J Clin Psychiatry. 1990 Dec;51 Suppl A:12-6. PMID 2258371
- [Background] Keller MB, Hanks DL. Course and outcome in panic disorder. Prog Neuropsychopharmacol Biol Psychiatry. 1993 Jul;17(4):551-70. doi: 10.1016/0278-5846(93)90005-d. PMID 8362071
- [Background] Roy-Byrne PP, Stang P, Wittchen HU, Ustun B, Walters EE, Kessler RC. Lifetime panic-depression comorbidity in the National Comorbidity Survey. Association with symptoms, impairment, course and help-seeking. Br J Psychiatry. 2000 Mar;176:229-35. doi: 10.1192/bjp.176.3.229. PMID 10755069
- [Background] Weissman MM, Klerman GL, Markowitz JS, Ouellette R. Suicidal ideation and suicide attempts in panic disorder and attacks. N Engl J Med. 1989 Nov 2;321(18):1209-14. doi: 10.1056/NEJM198911023211801. PMID 2797086
- [Background] Markowitz JS, Weissman MM, Ouellette R, Lish JD, Klerman GL. Quality of life in panic disorder. Arch Gen Psychiatry. 1989 Nov;46(11):984-92. doi: 10.1001/archpsyc.1989.01810110026004. PMID 2684086
- [Background] Sun H, Kennedy WP, Wilbraham D, Lewis N, Calder N, Li X, Ma J, Yee KL, Ermlich S, Mangin E, Lines C, Rosen L, Chodakewitz J, Murphy GM. Effects of suvorexant, an orexin receptor antagonist, on sleep parameters as measured by polysomnography in healthy men. Sleep. 2013 Feb 1;36(2):259-67. doi: 10.5665/sleep.2386. PMID 23372274
- [Background] Herring WJ, Snyder E, Budd K, Hutzelmann J, Snavely D, Liu K, Lines C, Roth T, Michelson D. Orexin receptor antagonism for treatment of insomnia: a randomized clinical trial of suvorexant. Neurology. 2012 Dec 4;79(23):2265-74. doi: 10.1212/WNL.0b013e31827688ee. Epub 2012 Nov 28. PMID 23197752
- [Background] Flores A, Valls-Comamala V, Costa G, Saravia R, Maldonado R, Berrendero F. The hypocretin/orexin system mediates the extinction of fear memories. Neuropsychopharmacology. 2014 Nov;39(12):2732-41. doi: 10.1038/npp.2014.146. Epub 2014 Jun 16. PMID 24930888
- [Background] Johnson PL, Samuels BC, Fitz SD, Lightman SL, Lowry CA, Shekhar A. Activation of the orexin 1 receptor is a critical component of CO2-mediated anxiety and hypertension but not bradycardia. Neuropsychopharmacology. 2012 Jul;37(8):1911-22. doi: 10.1038/npp.2012.38. Epub 2012 Mar 28. PMID 22453138
- [Background] Perna G, Battaglia M, Garberi A, Arancio C, Bertani A, Bellodi L. Carbon dioxide/oxygen challenge test in panic disorder. Psychiatry Res. 1994 May;52(2):159-71. doi: 10.1016/0165-1781(94)90085-x. PMID 7972572
- [Background] Williams RH, Jensen LT, Verkhratsky A, Fugger L, Burdakov D. Control of hypothalamic orexin neurons by acid and CO2. Proc Natl Acad Sci U S A. 2007 Jun 19;104(25):10685-90. doi: 10.1073/pnas.0702676104. Epub 2007 Jun 11. PMID 17563364
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Brundin L, Bjorkqvist M, Petersen A, Traskman-Bendz L. Reduced orexin levels in the cerebrospinal fluid of suicidal patients with major depressive disorder. Eur Neuropsychopharmacol. 2007 Sep;17(9):573-9. doi: 10.1016/j.euroneuro.2007.01.005. Epub 2007 Mar 7. PMID 17346943
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Mignot E, Lammers GJ, Ripley B, Okun M, Nevsimalova S, Overeem S, Vankova J, Black J, Harsh J, Bassetti C, Schrader H, Nishino S. The role of cerebrospinal fluid hypocretin measurement in the diagnosis of narcolepsy and other hypersomnias. Arch Neurol. 2002 Oct;59(10):1553-62. doi: 10.1001/archneur.59.10.1553. PMID 12374492
- [Background] Shear MK, Brown TA, Barlow DH, Money R, Sholomskas DE, Woods SW, Gorman JM, Papp LA. Multicenter collaborative panic disorder severity scale. Am J Psychiatry. 1997 Nov;154(11):1571-5. doi: 10.1176/ajp.154.11.1571. PMID 9356566
- [Background] Goddard AW, Woods SW, Sholomskas DE, Goodman WK, Charney DS, Heninger GR. Effects of the serotonin reuptake inhibitor fluvoxamine on yohimbine-induced anxiety in panic disorder. Psychiatry Res. 1993 Aug;48(2):119-33. doi: 10.1016/0165-1781(93)90036-g. PMID 8416022
- [Background] Thompson JP, Watt P, Sanghavi S, Strupish JW, Lambert DG. A comparison of cerebrospinal fluid and plasma urotensin II concentrations in normotensive and hypertensive patients undergoing urological surgery during spinal anesthesia: a pilot study. Anesth Analg. 2003 Nov;97(5):1501-1503. doi: 10.1213/01.ANE.0000086723.97421.BC. PMID 14570674

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Per IRB records, 3 participants enrolled and 2 completed the study. PI left institution and all efforts to locate data have been exhausted.
Groups:
- Suvorexant Group: In this arm, subjects will receive 10 mg suvorexant 2 hours before a one-minute 35% CO2 challenge.
  suvorexant
- Placebo Group: In this arm, subjects will receive a placebo, compounded to look identical to the study drug, 2 hours before a one-minute 35% CO2 challenge.
  placebo
Period: Overall Study
Arm/Group | Suvorexant Group | Placebo Group
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: PI left institution and all efforts to locate data have been exhausted.
Groups:
- Total: Total of all reporting groups
Arm/Group | Suvorexant Group | Placebo Group | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Change in Orexin Levels (Blood) +1 Minute
Description: Change in orexin levels from baseline to +1 min post-CO2 challenge
Time Frame: Baseline and +1 minute post-CO2 challenge
Population: PI left institution and all efforts to locate data have been exhausted.
Arm/Group | Suvorexant Group | Placebo Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Orexin Levels (Blood) +5 Minutes
Description: Change in orexin levels from baseline to +5 min post-CO2 challenge
Time Frame: Baseline and +5 minutes post-CO2 challenge
Population: PI left institution and all efforts to locate data have been exhausted.
Arm/Group | Suvorexant Group | Placebo Group
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change in Orexin Levels (Blood) +15 Minutes
Description: Change in orexin levels from baseline to +15 min post-CO2 challenge
Time Frame: Baseline and +15 minutes post-CO2 challenge
Population: PI left institution and all efforts to locate data have been exhausted.
Arm/Group | Suvorexant Group | Placebo Group
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Change in Orexin Levels (Blood) +60 Minutes
Description: Change in orexin levels from baseline to +60 min post-CO2 challenge
Time Frame: Baseline and +60 minutes post-CO2 challenge
Population: PI left institution and all efforts to locate data have been exhausted.
Arm/Group | Suvorexant Group | Placebo Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: PI left institution and all efforts to locate data have been exhausted.
Description: PI left institution and all efforts to locate data have been exhausted.
Arm/Group | Suvorexant Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT02593682/Prot_SAP_000.pdf